CLINICAL TRIAL: NCT05427253
Title: A Double-blind, Placebo-controlled, Randomised, First in Human Trial to Evaluate the Safety, Tolerability and Pharmacokinetics of Single and Multiple Ascending Oral Doses of C106 in Healthy Male and Female Subjects
Brief Title: First-in-human Trial to Evaluate the Safety, Tolerability and Pharmacokinetics of C106 in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Vicore Pharma AB (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: VP-C106-101
Record Dates: First submitted 2022-06-07; First posted 2022-06-22 (Actual); Results first posted 2025-01-31 (Actual); Last update posted 2025-01-31 (Actual); Status verified 2024-12

CONDITIONS: Safety Issues; Tolerance; Idiopathic Pulmonary Fibrosis; Pulmonary Hypertension
MeSH Terms: conditions — Idiopathic Pulmonary Fibrosis; Hypertension, Pulmonary

STUDY DESIGN:
Intervention Model Description: Part A, single ascending dose (SAD) including a food interaction cohort Part B, multiple ascending dose (MAD)
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The IMP, i.e., the C106 and the placebo oral solutions, are identical in appearance. Both solutions are colourless to yellow. Hence, it is expected that the subjects, Investigator and other site personnel will remain unaware of treatment allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- C106 solution (Experimental): Part A: Oral administration start dose, Single dose 5 mg Part B: Oral administration start dose 20 mg twice daily for 8 days
  Interventions: Drug: C106 solution
- Placebo (Placebo Comparator): Part A and B: Placebo to C106 without the active pharmaceutical ingredient
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: C106 solution — selective nonpeptide angiotensin II type 2 receptor (AT2R) agonist
  Arms: C106 solution
Drug: Placebo — Placebo for C106 solution
  Arms: Placebo

SUMMARY:
This is a FIH, double-blind, placebo-controlled, within-group randomised, trial designed to evaluate the safety, tolerability, and pharmacokinetics (PK) of single and multiple ascending oral doses of compound 106 (C106) in healthy females of non-childbearing potential and healthy males.

The trial will be conducted in 2 parts:

Part A, single ascending dose (SAD) including a food interaction cohort: safety, tolerability, and PK in healthy males and healthy females of non-childbearing potential receiving single ascending doses of C106.

Part B, multiple ascending dose (MAD): safety, tolerability, and PK in healthy males and healthy females of non-childbearing potential receiving twice daily multiple ascending doses of C106 for 8 days.

ELIGIBILITY:
Inclusion Criteria:

1. Willing and able to give written informed consent for participation in the trial.
2. Healthy males and females of non-childbearing potential aged 18-65 years inclusive.
3. Body Mass Index (BMI) ≥ 18.5 and ≤ 30.0 kg/m2
4. Clinically normal medical history, physical findings, vital signs, ECG, and laboratory values at the time of screening, as judged by the Investigator
5. Women of non-childbearing potential, defined as pre-menopausal females who are sterilized (tubal ligation or permanent bilateral occlusion of fallopian tubes); or females who have undergone hysterectomy or bilateral oophorectomy; or post-menopausal defined as 12 months of amenorrhea (in questionable cases a blood sample with simultaneous detection of follicle stimulating hormone [FSH] ≥ 25 IU/L is confirmatory).

Male subjects must be willing to use condom or be vasectomised or practice sexual abstinence to prevent pregnancy and drug exposure of a partner and refrain from donating sperm from the date of dosing until 3 months after (last) dosing with the IMP. Their female partner of child-bearing potential must use highly effective contraceptive methods with a failure rate of < 1% to prevent pregnancy (combined [oestrogen and progestogen containing] hormonal contraception associated with inhibition of ovulation [oral, intravaginal, transdermal], progestogen-only hormonal contraception associated with inhibition of ovulation [oral, injectable, implantable], intrauterine device [IUD]or intrauterine hormone-releasing system [IUS]) from at least 4 weeks prior to dose to 3 months after last dose.

Exclusion Criteria:

1. History of any clinically significant disease or disorder which, in the opinion of the Investigator, may either put the subject at risk because of participation in the trial, or influence the results or the subject's ability to participate in the trial.
2. Any clinically significant illness, medical/surgical procedure, or trauma within 4 weeks of the first administration of IMP.
3. Malignancy within the past 5 years except for in situ removal of basal cell carcinoma.
4. Any planned major surgery within the duration of the trial.
5. Any positive result on screening for serum hepatitis B surface antigen, hepatitis C antibody and Human Immunodeficiency Virus (HIV).
6. After 10 minutes supine rest at the time of screening, any vital signs values outside the following ranges:

   * Systolic blood pressure <90 or >140 mmHg, or
   * Diastolic blood pressure <50 or >90 mmHg, or
   * Pulse <40 or >90 bpm
7. Prolonged QTcF (>450 ms), PR interval < 120 ms or > 240 ms, QRS>115 ms, clinically significant cardiac arrhythmias or any clinically significant abnormalities in the resting ECG at the time of screening, as judged by the Investigator.
8. History of severe allergy/hypersensitivity or ongoing allergy/hypersensitivity, as judged by the Investigator, or history of hypersensitivity to drugs with a similar chemical structure or class to C106.
9. Regular use of any prescribed or non-prescribed medication including antacids, analgesics, herbal remedies, vitamins and minerals within 2 weeks prior to the (first) administration of IMP, at the discretion of the Investigator.
10. Planned treatment or treatment with another investigational drug within 3 months prior to Day -1. Subjects consented and screened but not dosed in previous clinical trials are not excluded.
11. Current smokers or users of nicotine products. Irregular use of nicotine (e.g., smoking, snuffing, chewing tobacco) less than three times per week is allowed before screening visit.
12. Positive screen for drugs of abuse or alcohol at screening or on admission to the unit prior to administration of the IMP.
13. History of alcohol abuse or excessive intake of alcohol, as judged by the Investigator.
14. Presence or history of drug abuse, as judged by the Investigator.
15. History of, or current use of, anabolic steroids.
16. Excessive caffeine consumption defined by a daily intake of >5 cups of caffeine containing beverages.
17. Plasma donation within one month of screening or blood donation (or corresponding blood loss) during the three months prior to screening.
18. Investigator considers the subject unlikely to comply with trial procedures, restrictions, and requirements.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2022-06-08 (Actual); Primary Completion 2023-06-22 (Actual); Study Completion 2023-06-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Måns Jergil, PhD, Study Director — CTC Clinical Trial Consultants AB (CTC); Helena Litorp, MD, PhD, Principal Investigator — CTC Clinical Trial Consultants AB (CTC)
Locations (1):
- CTC Clinical Trial Consultants AB, Uppsala, Sweden

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The subjects were recruited from CTC's database of healthy volunteers and patients, as well as from strategic marketing campaigns. Advertisements in social media and other media.
  Single ascending dose (SAD) part: First subject screened: 08-Jun-2022 Last subject completed: 09-May-2023 Multiple ascending dose (MAD) part: First subject screened: 19-Aug-2022 Last subject completed: 22-Jun-2023
Pre-assignment Details: SAD part: Screened - 92 subjects, included - 48 subjects. Subjects in the SAD Part Cohort 4, dose 180 mg group were supposed to completed additional trial visits exploring single dose administration of C106 under fed conditions, this group is called SAD Part Cohort 4, dose 180 mg fasted first, then Dose 180 mg Fed.
  MAD part: Screened - 77 subjects, included 32 subjects. 28 subjects completed all 3 trial visits (multiple dose administration of C106). 4 subjects were withdrawn from the trial.
Groups:
- SAD Part Cohort 1, Dose 5 mg: Oral administration, Single dose 5 mg oral solution
  C106 solution: selective nonpeptide angiotensin II type 2 receptor (AT2R) agonist
- SAD Part Cohort 2, Dose 30 mg: Oral administration, Single dose 30 mg oral solution
  C106 solution: selective nonpeptide angiotensin II type 2 receptor (AT2R) agonist
- SAD Part Cohort 3, Dose 60 mg: Oral administration, Single dose 60 mg oral solution
  C106 solution: selective nonpeptide angiotensin II type 2 receptor (AT2R) agonist
- SAD Part Cohort 4, Dose 180 mg Fasted First, Then Dose 180 mg Fed: Oral administration, Single dose 180 mg oral solution
  Subjects proceed from the SAD Part Cohort 4, dose 180 mg fasting after a washout period of at least 5 half-lives of C106 to a second period where the intervention of 180 mg is given under fed condition.
  C106 solution: selective nonpeptide angiotensin II type 2 receptor (AT2R) agonist
- SAD Part Cohort 5, Dose 240 mg: Oral administration, Single dose 240 mg oral solution
  C106 solution: selective nonpeptide angiotensin II type 2 receptor (AT2R) agonist
- SAD Part, Cohort 6, Dose 300 mg: Oral administration, Single dose 300 mg oral solution
  C106 solution: selective nonpeptide angiotensin II type 2 receptor (AT2R) agonist
- SAD Part, Placebo: Oral administration, Single dose placebo oral solution
- MAD Part, Dose 40mg: Oral administration dose 40 mg twice daily for 8 days
  C106 solution: selective nonpeptide angiotensin II type 2 receptor (AT2R) agonist
- MAD Part, Dose 100mg: Oral administration dose 100 mg twice daily for 8 days
  C106 solution: selective nonpeptide angiotensin II type 2 receptor (AT2R) agonist
- MAD Part, Dose 140mg: Oral administration dose 140 mg twice daily for 8 days
  C106 solution: selective nonpeptide angiotensin II type 2 receptor (AT2R) agonist
- MAD Part, Dose 180mg: Oral administration dose 180 mg twice daily for 8 days
  C106 solution: selective nonpeptide angiotensin II type 2 receptor (AT2R) agonist
- MAD Part, Placebo: Oral administration of placebo oral solution twice daily for 8 days
Period: Intervention Under Fasting Condition
Arm/Group | SAD Part Cohort 1, Dose 5 mg | SAD Part Cohort 2, Dose 30 mg | SAD Part Cohort 3, Dose 60 mg | SAD Part Cohort 4, Dose 180 mg Fasted First, Then Dose 180 mg Fed | SAD Part Cohort 5, Dose 240 mg | SAD Part, Cohort 6, Dose 300 mg | SAD Part, Placebo | MAD Part, Dose 40mg | MAD Part, Dose 100mg | MAD Part, Dose 140mg | MAD Part, Dose 180mg | MAD Part, Placebo
Started | 6 | 6 | 6 | 6 | 6 | 6 | 12 | 6 | 6 | 6 | 6 | 8
Completed | 6 | 6 | 6 | 6 | 6 | 6 | 12 | 6 | 4 | 6 | 4 | 8
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 2 | 0
Period: Wash Out for SAD Part Cohort 4, Dose 180
Arm/Group | SAD Part Cohort 1, Dose 5 mg | SAD Part Cohort 2, Dose 30 mg | SAD Part Cohort 3, Dose 60 mg | SAD Part Cohort 4, Dose 180 mg Fasted First, Then Dose 180 mg Fed | SAD Part Cohort 5, Dose 240 mg | SAD Part, Cohort 6, Dose 300 mg | SAD Part, Placebo | MAD Part, Dose 40mg | MAD Part, Dose 100mg | MAD Part, Dose 140mg | MAD Part, Dose 180mg | MAD Part, Placebo
Started | 0 | 0 | 0 | 6 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 6 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Intervention Under Fed Condition
Arm/Group | SAD Part Cohort 1, Dose 5 mg | SAD Part Cohort 2, Dose 30 mg | SAD Part Cohort 3, Dose 60 mg | SAD Part Cohort 4, Dose 180 mg Fasted First, Then Dose 180 mg Fed | SAD Part Cohort 5, Dose 240 mg | SAD Part, Cohort 6, Dose 300 mg | SAD Part, Placebo | MAD Part, Dose 40mg | MAD Part, Dose 100mg | MAD Part, Dose 140mg | MAD Part, Dose 180mg | MAD Part, Placebo
Started | 0 | 0 | 0 | 5 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 5 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- SAD Part Cohort 4, Dose 180 mg, Fasted First, Then Dose 180 mg Fed: Oral administration, Single dose 180 mg oral solution, Fasted First, Then Dose 180 mg Fed
  C106 solution: selective nonpeptide angiotensin II type 2 receptor (AT2R) agonist
- Total: Total of all reporting groups
Arm/Group | SAD Part Cohort 1, Dose 5 mg | SAD Part Cohort 2, Dose 30 mg | SAD Part Cohort 3, Dose 60 mg | SAD Part Cohort 4, Dose 180 mg, Fasted First, Then Dose 180 mg Fed | SAD Part Cohort 5, Dose 240 mg | SAD Part, Cohort 6, Dose 300 mg | SAD Part, Placebo | MAD Part, Dose 40mg | MAD Part, Dose 100mg | MAD Part, Dose 140mg | MAD Part, Dose 180mg | MAD Part, Placebo | Total
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 12 | 6 | 6 | 6 | 6 | 8 | 80
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 6 | 6 | 6 | 6 | 6 | 6 | 12 | 6 | 6 | 6 | 6 | 8 | 80
  >=65 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.5 (11.7) | 47.2 (12.9) | 35.0 (9.4) | 40.2 (16.2) | 38.7 (14.0) | 50.8 (17.0) | 46.5 (14.4) | 39.3 (10.6) | 29.0 (5.3) | 31.3 (7.1) | 37.2 (9.9) | 36.6 (13.0) | 39.7 (13.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 1 | 0 | 1 | 1 | 4 | 3 | 1 | 0 | 1 | 1 | 1 | 14
  Male | 6 | 5 | 6 | 5 | 5 | 2 | 9 | 5 | 6 | 5 | 5 | 7 | 66
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
  White | 6 | 5 | 6 | 6 | 6 | 6 | 11 | 6 | 6 | 4 | 5 | 8 | 75
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Sweden | 6 | 6 | 6 | 6 | 6 | 6 | 12 | 6 | 6 | 6 | 6 | 8 | 80

OUTCOME MEASURES:

1. Primary Outcome: Total Number of Treatment Emergent Adverse Events (AEs) and Serious AEs (SAEs)
Description: AE reporting and questioning. AEs must be recorded in the AE Log of the eCRF. The Investigator must provide information on the AE, preferably with a diagnosis or at least with signs and symptoms; start and stop dates, start and stop time; intensity; causal relationship to IMP; action taken, and outcome.
  If the AE is serious, this must be indicated in the eCRF. AEs, including out-of-range clinically significant clinical safety laboratory values, must be recorded individually, except when considered manifestations of the same medical condition or disease state; in such cases, they must be recorded under a single diagnosis.
  The grading of the severity/intensity (grade 1 to grade 5) of AEs followed the common terminology criteria for AEs (CTCAE) v5.0. The causal relationship between AEs and the IMP was assessed as related, not related or not applicable.
Time Frame: From date of signing informed consent until End of Study, assessed up to Day 22
Population: SAD: The withdrawn subject was part of Cohort 4 fed condition. .The subject was excluded from the trial before completing the food interaction visit.
  MAD: Two (2) subjects in the 100 mg C106 dose group had AEs (common cold) that lead to subject withdrawal from the trial.
Measure: Number; unit: Number of events
Groups:
- SAD Part Cohort 4, Dose 180 mg: Oral administration, Single dose 180 mg oral solution
  C106 solution: selective nonpeptide angiotensin II type 2 receptor (AT2R) agonist
- SAD Part Cohort 4, Dose 180 mg Fed: Oral administration, Single dose 180 mg oral solution in fed condition.
  C106 solution: selective nonpeptide angiotensin II type 2 receptor (AT2R) agonist
Arm/Group | SAD Part Cohort 1, Dose 5 mg | SAD Part Cohort 2, Dose 30 mg | SAD Part Cohort 3, Dose 60 mg | SAD Part Cohort 4, Dose 180 mg | SAD Part Cohort 4, Dose 180 mg Fed | SAD Part Cohort 5, Dose 240 mg | SAD Part, Cohort 6, Dose 300 mg | SAD Part, Placebo | MAD Part, Dose 40mg | MAD Part, Dose 100mg | MAD Part, Dose 140mg | MAD Part, Dose 180mg | MAD Part, Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 5 | 6 | 6 | 12 | 6 | 6 | 6 | 6 | 8
Number of events
  Adverse events | 5 | 5 | 3 | 2 | 2 | 7 | 8 | 4 | 11 | 10 | 15 | 7 | 21
  Serious Adverse events | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

2. Primary Outcome: Number of Reported Clinically Significant Changes From Baseline in 12-lead Electrocardiograms (ECGs)
Description: Single 12-lead ECG will be recorded in supine position after 10 minutes of rest using an ECG machine. Abnormalities will be specified and documented as clinically significant or not clinically significant.
  Heart rate (HR) and PR, QRS, QT, and QTcF intervals were recorded.
Time Frame: Part A: Up to Day 10. Part B: Up to Day 22.
Population: Data were presented using summary statistics..
Measure: Number; unit: Number of events
Arm/Group | SAD Part Cohort 1, Dose 5 mg | SAD Part Cohort 2, Dose 30 mg | SAD Part Cohort 3, Dose 60 mg | SAD Part Cohort 4, Dose 180 mg | SAD Part Cohort 4, Dose 180 mg Fed | SAD Part Cohort 5, Dose 240 mg | SAD Part, Cohort 6, Dose 300 mg | SAD Part, Placebo | MAD Part, Dose 40mg | MAD Part, Dose 100mg | MAD Part, Dose 140mg | MAD Part, Dose 180mg | MAD Part, Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 5 | 6 | 6 | 12 | 6 | 6 | 6 | 6 | 8
Number of events | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0

3. Primary Outcome: Number of Reported Clinically Significant Changes in Vital Signs
Description: Systolic and diastolic blood pressure and pulse were measured in supine position after 10 minutes of rest. The respiratory rate was assessed. Body temperature was measured using a digital thermometer on Day -1 of each part.
Time Frame: Part A: Up to Day 3, Part B: Up to Day 10. Vital signs were measured at pre-defined timepoints during the trial.
Population: Data were presented using summary statistics.
Measure: Number; unit: Number of events
Arm/Group | SAD Part Cohort 1, Dose 5 mg | SAD Part Cohort 2, Dose 30 mg | SAD Part Cohort 3, Dose 60 mg | SAD Part Cohort 4, Dose 180 mg | SAD Part Cohort 4, Dose 180 mg Fed | SAD Part Cohort 5, Dose 240 mg | SAD Part, Cohort 6, Dose 300 mg | SAD Part, Placebo | MAD Part, Dose 40mg | MAD Part, Dose 100mg | MAD Part, Dose 140mg | MAD Part, Dose 180mg | MAD Part, Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 5 | 6 | 6 | 12 | 6 | 6 | 6 | 6 | 8
Number of events
  Blood pressure | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 0
  Pulse | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Respiratory rate | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 1 | 2

4. Primary Outcome: Number of Clinically Significant Changes in Laboratory Safety Variables (Haematology, Coagulation, Clinical Chemistry and Urine Analysis)
Description: Blood samples for analysis of clinical chemistry, haematology, and coagulation parameters were collected through venepuncture or an indwelling venous catheter.
Time Frame: Part A: Up to Day 3, Part B: Up to Day 10. Safety laboratory samples were collected at pre-defined timepoints during the trial.
Population: Data were presented using summary statistics.
Measure: Number; unit: Number of events
Arm/Group | SAD Part Cohort 1, Dose 5 mg | SAD Part Cohort 2, Dose 30 mg | SAD Part Cohort 3, Dose 60 mg | SAD Part Cohort 4, Dose 180 mg | SAD Part Cohort 4, Dose 180 mg Fed | SAD Part Cohort 5, Dose 240 mg | SAD Part, Cohort 6, Dose 300 mg | SAD Part, Placebo | MAD Part, Dose 40mg | MAD Part, Dose 100mg | MAD Part, Dose 140mg | MAD Part, Dose 180mg | MAD Part, Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 5 | 6 | 6 | 12 | 6 | 6 | 6 | 6 | 8
Number of events
  Clinical chemistry | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Haematology | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Coagulation | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Urinalysis | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

5. Primary Outcome: Number of Reported Clinically Significant Changes in Physical Examinations.
Description: Any abnormalities will be specified and documented as clinically significant or not clinically significant. Abnormal findings assessed as clinically significant will be reported as AEs.
  A complete physical examination will include assessments of the head, eyes, ears, nose, throat, skin, neurological, lungs, cardiovascular, and abdomen.
  .
Time Frame: Physical examination was performed at pre-defined timepoints during the trial. Part A: Day 7, Part B: Day 22
Population: Data were presented using summary statistics.
Measure: Number; unit: Number of events
Arm/Group | SAD Part Cohort 1, Dose 5 mg | SAD Part Cohort 2, Dose 30 mg | SAD Part Cohort 3, Dose 60 mg | SAD Part Cohort 4, Dose 180 mg | SAD Part Cohort 4, Dose 180 mg Fed | SAD Part Cohort 5, Dose 240 mg | SAD Part, Cohort 6, Dose 300 mg | SAD Part, Placebo | MAD Part, Dose 40mg | MAD Part, Dose 100mg | MAD Part, Dose 140mg | MAD Part, Dose 180mg | MAD Part, Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 5 | 6 | 6 | 12 | 6 | 6 | 6 | 6 | 8
Number of events | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: AEs (including serious AEs [SAEs]) were collected from the signing of the informed consent form until the end-of-trial visit for each subject, ranging from up to 37 days in SAD part to up to 47 days in MAD part.
Description: The grading of the severity/intensity (grade 1 to grade 5) of AEs followed the common terminology criteria for AEs (CTCAE) v5.0. The causal relationship between AEs and the IMP was assessed as related, not related or not applicable.
Arm/Group | SAD Part Cohort 1, Dose 5 mg | SAD Part Cohort 2, Dose 30 mg | SAD Part Cohort 3, Dose 60 mg | SAD Part Cohort 4, Dose 180 mg | SAD Part Cohort 4, Dose 180 mg Fed | SAD Part Cohort 5, Dose 240 mg | SAD Part, Cohort 6, Dose 300 mg | SAD Part, Placebo | MAD Part, Dose 40mg | MAD Part, Dose 100mg | MAD Part, Dose 140mg | MAD Part, Dose 180mg | MAD Part, Placebo
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/6 | 0/6 | 0/6 | 0/5 | 0/6 | 0/6 | 0/12 | 0/6 | 0/6 | 0/6 | 0/6 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/6 | 0/6 | 0/6 | 0/5 | 0/6 | 0/6 | 0/12 | 0/6 | 0/6 | 0/6 | 0/6 | 0/8
Other Adverse Events (participants affected / at risk) | 2/6 | 2/6 | 2/6 | 2/6 | 2/5 | 2/6 | 4/6 | 4/12 | 4/6 | 5/6 | 5/6 | 4/6 | 8/8
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SAD Part Cohort 1, Dose 5 mg (N=6) | SAD Part Cohort 2, Dose 30 mg (N=6) | SAD Part Cohort 3, Dose 60 mg (N=6) | SAD Part Cohort 4, Dose 180 mg (N=6) | SAD Part Cohort 4, Dose 180 mg Fed (N=5) | SAD Part Cohort 5, Dose 240 mg (N=6) | SAD Part, Cohort 6, Dose 300 mg (N=6) | SAD Part, Placebo (N=12) | MAD Part, Dose 40mg (N=6) | MAD Part, Dose 100mg (N=6) | MAD Part, Dose 140mg (N=6) | MAD Part, Dose 180mg (N=6) | MAD Part, Placebo (N=8)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (3) | 0 (0) | 1 (1) | 3 (5) | 1 (4) | 1 (1) | 4 (5)
Paraesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Restless legs syndrome (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dysgeusia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypoesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Fatigue (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Malaise (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Swelling (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Chest discomfort (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Feeling hot (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Flatulence (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (3)
Hypoaesthesia oral (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthropod sting (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vascular access site inflammation (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Skin burning sensation (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Onychoclasis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Atrioventricular block second degree (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bradycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Atrioventricular block first degree (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rhinitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tooth infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Blood pressure increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Respiratory rate decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 2 (2)
Blepharospasm (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eye paraesthesia (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Groin pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Irritability (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nasal pruritus (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oropharyngeal discomfort (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bladder pain (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urinary incontinence (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-02-27): https://cdn.clinicaltrials.gov/large-docs/53/NCT05427253/Prot_SAP_000.pdf